CLINICAL TRIAL: NCT02612688
Title: PROVEN: Pragmatic Trial of Video Education in Nursing Homes
Brief Title: Pragmatic Trial of Video Education in Nursing Homes
Acronym: PROVEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Hebrew SeniorLife (Other); Massachusetts General Hospital (Other); Genesis HealthCare (Other); PruittHealth (Other)
Responsible Party: Principal Investigator, Vincent Mor, Professor of Medical Science, Florence Pirce Grant University Professor, Health Services, Policy & Practice, Brown University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 4UH3AG049619-02 (NIH); 4UH3AG049619-02 (NIH)
Record Dates: First submitted 2015-11-19; First posted 2015-11-24 (Estimated); Results first posted 2020-06-18 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-09

CONDITIONS: Alzheimer Disease; Dementia; Heart Failure; Pulmonary Disease, Chronic Obstructive
Keywords: Advance Care Planning; Advance Directives; Alzheimer Disease; Dementia; Do-Not-Resuscitate Orders; Enteral Nutrition; Heart Failure; Hospices; Hospitalization; Instructional Films and Videos; Intubation; Nursing Homes; Parenteral Nutrition; Pragmatic Clinical Trials; Pulmonary Disease, Chronic Obstructive; Randomized Controlled Trials; Resuscitation Orders; Skilled Nursing Facilities
MeSH Terms: conditions — Alzheimer Disease; Dementia; Heart Failure; Pulmonary Disease, Chronic Obstructive; Hyperphagia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACP Video Program (Experimental): Facility asked to implement ACP Video Program
  Interventions: Behavioral: ACP Video Program
- Usual ACP procedures (No Intervention): Facility follows usual ACP procedures

INTERVENTIONS:
Behavioral: ACP Video Program — The ACP Video Program consists of five videos that address ACP decisions: (1) General Goals of Care, (2) Goals of Care for Advanced Dementia, (3) Hospice, (4) Hospitalization, and (5) ACP for Healthy Patients. NH staff will offer videos to patients at these clinical triggers: (1) Within 7 days of admission or readmission; (2) Every 6 months for long-stay patients; (3) When there is a significant change in clinical status; (4) When a treatment decision arises for which there is a specific video; and (5) Special circumstances when goals of care are being considered (e.g., family visiting).
  Arms: ACP Video Program

SUMMARY:
This is a pragmatic cluster-randomized control trial (RCT) of an Advance Care Planning (ACP) Video Program for nursing home (NH) patients ≥ 65 years old who are cared for in 360 NH facilities (intervention arm n=119; control arm n=241) within two NH health care systems: Genesis HealthCare and PruittHealth. The intervention NH facilities will implement the ACP Video Program, while the control NH facilities will follow their usual ACP procedures. The trial will evaluate the effectiveness of the ACP Video Program by comparing hospitalizations, advance directives, and hospice use in the intervention vs. control NHs.

DETAILED DESCRIPTION:
Nursing homes are complex health care systems that serve increasingly sick patients who have advanced comorbid conditions. NHs are often charged with guiding patients through decisions about the direction of their treatment. Patients at NHs commonly get aggressive care that may be inconsistent with their preferences and of little clinical benefit. Identifying effective approaches that NHs can use to better promote goal-directed care and optimize resources is a research, public health, and clinical priority.

Advance care planning is the most consistent modifiable factor associated with better palliative care outcomes. Traditional ACP relies on verbal descriptions of hypothetical health states and treatments. This approach is limited because complex scenarios are difficult to envision, counseling is inconsistent, and verbal explanations are hindered by literacy and language barriers.

To address these shortcomings, the PROVEN project has developed video-assisted ACP decision-support tools that have shown efficacy in small randomized controlled trials. While several large health care systems have begun to adopt the videos, efforts have not rigorously evaluated outcomes-a critical step prior to widespread implementation.

The goal of PROVEN is to conduct a pragmatic cluster-randomized trial to evaluate the effectiveness of the ACP Video Program in the NH setting by partnering with 2 large health care systems that operate 456 nursing homes nationwide. This work has the potential to improve the care provided to millions of older Americans in nursing homes and enable future pragmatic trials in this setting.

ELIGIBILITY:
Inclusion Criteria:

* Facilities are within Genesis HealthCare or PruittHealth health care systems
* Facilities have facility identifiers that indicate that they are Medicare/Medicaid-certified nursing facilities in the U.S.
* Facilities serve both short and long-stay patients
* Facilities have >50 beds
* Facilities have an electronic medical records system
* Facilities had at least 20 admissions and 20 annual Minimum Data Set (MDS) assessments (regardless of whether they were discharged alive) in 2013

Exclusion Criteria:

* Facilities excluded per corporate leaders in health care system because of recent turnover in NH administrator or Director of Nursing
* Facilities excluded per corporate leaders in health care system because of recent bad state or federal quality assurance survey (e.g. restriction on admissions, levied large civil monetary penalty, etc.)
* Facilities excluded per corporate leaders in health care system because of current new initiatives/competing demands

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 197692 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Mor, PhD, Principal Investigator — Brown University; Susan Mitchell, MD, MPH, Principal Investigator — Hebrew SeniorLife; Angelo Volandes, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - PruittHealth, Norcross, Georgia
  - Genesis HealthCare, Kennett Square, Pennsylvania

REFERENCES:
- [Derived] McCreedy EM, Yang X, Mitchell SL, Gutman R, Teno J, Loomer L, Moyo P, Volandes A, Gozalo PL, Belanger E, Ogarek J, Mor V. Effect of advance care planning video on do-not-hospitalize orders for nursing home residents with advanced illness. BMC Geriatr. 2022 Apr 8;22(1):298. doi: 10.1186/s12877-022-02970-3. PMID 35392827
- [Derived] Mitchell SL, Volandes AE, Gutman R, Gozalo PL, Ogarek JA, Loomer L, McCreedy EM, Zhai R, Mor V. Advance Care Planning Video Intervention Among Long-Stay Nursing Home Residents: A Pragmatic Cluster Randomized Clinical Trial. JAMA Intern Med. 2020 Aug 1;180(8):1070-1078. doi: 10.1001/jamainternmed.2020.2366. PMID 32628258
- [Derived] Palmer JA, Parker VA, Barre LR, Mor V, Volandes AE, Belanger E, Loomer L, McCreedy E, Mitchell SL. Understanding implementation fidelity in a pragmatic randomized clinical trial in the nursing home setting:a mixed-methods examination. Trials. 2019 Nov 28;20(1):656. doi: 10.1186/s13063-019-3725-5. PMID 31779684
- [Derived] Palmer JA, Parker VA, Mor V, Volandes AE, Barre LR, Belanger E, Carter P, Loomer L, McCreedy E, Mitchell SL. Barriers and facilitators to implementing a pragmatic trial to improve advance care planning in the nursing home setting. BMC Health Serv Res. 2019 Jul 29;19(1):527. doi: 10.1186/s12913-019-4309-5. PMID 31357993
- [Derived] Loomer L, McCreedy E, Belanger E, Palmer JA, Mitchell SL, Volandes AE, Mor V. Nursing Home Characteristics Associated With Implementation of an Advance Care Planning Video Intervention. J Am Med Dir Assoc. 2019 Jul;20(7):804-809.e1. doi: 10.1016/j.jamda.2019.01.133. Epub 2019 Mar 7. PMID 30852167
- [Derived] Palmer JA, Mor V, Volandes AE, McCreedy E, Loomer L, Carter P, Dvorchak F, Mitchell SL. A dynamic application of PRECIS-2 to evaluate implementation in a pragmatic, cluster randomized clinical trial in two nursing home systems. Trials. 2018 Aug 22;19(1):453. doi: 10.1186/s13063-018-2817-y. PMID 30134976
- See also: NIH Collaboratory website for UH3 Project: Pragmatic Trial of Video Education in Nursing Homes (PROVEN) — http://www.rethinkingclinicaltrials.org/uh3-project-pragmatic-trial-of-video-education-in-nursing-homes-proven/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ACP Video Program | Usual ACP Procedures
Started | 33035 | 70013
Completed | 33035 | 70013
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Advance Care Planning (ACP) Video Program: Facility asked to implement Advance Care Planning (ACP) Video Program
  ACP Video Program: The ACP Video Program consists of five videos that address ACP decisions: (1) General Goals of Care, (2) Goals of Care for Advanced Dementia, (3) Hospice, (4) Hospitalization, and (5) ACP for Healthy Patients. NH staff will offer videos to patients at these clinical triggers: (1) Within 7 days of admission or readmission; (2) Every 6 months for long-stay patients; (3) When there is a significant change in clinical status; (4) When a treatment decision arises for which there is a specific video; and (5) Special circumstances when goals of care are being considered (e.g., family visiting).
- Usual Advance Care Planning (ACP) Procedures: Facility follows usual Advance Care Planning (ACP) procedures
- Total: Total of all reporting groups
Arm/Group | Advance Care Planning (ACP) Video Program | Usual Advance Care Planning (ACP) Procedures | Total
Number analyzed (Participants) | 33035 | 70013 | 103048
Age, Continuous [Mean (Standard Deviation); unit: years] | 80.8 (8.9) | 80.9 (8.8) | 80.9 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19818 | 42170 | 61988
  Male | 13217 | 27843 | 41060
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 26888 | 58872 | 85760
  Race/Ethnicity: Black | 4904 | 8575 | 13479
  Race/Ethnicity: Asian | 240 | 617 | 857
  Race/Ethnicity: Hispanic | 287 | 626 | 913
  Race/Ethnicity: North American Native | 331 | 407 | 738
  Race/Ethnicity: Other | 215 | 491 | 706
  Race/Ethnicity: Unknown | 170 | 425 | 595

OUTCOME MEASURES:

1. Primary Outcome: Hospital Transfer Rate in Target Cohort
Description: Number of hospital transfers (number of transfers/person-days alive) over a 12-month observation period among Medicare fee-for-service long-stay residents (in a NH >=90 days) who are >=65 years old and who have EITHER advanced dementia or advanced congestive heart failure/chronic obstructive lung disease
Time Frame: 12-month observation period
Measure: Mean (Standard Deviation); unit: person-years
Arm/Group | ACP Video Program | Usual ACP Procedures
Number analyzed (Participants) | 4171 | 8308
person-years | 2.4 (11.8) | 2.8 (13.7)

2. Secondary Outcome: Hospital Transfer Rate Among Long-stay Residents Without Advanced Illness
Description: Number of hospital transfers (number of transfers/person-days alive) over a 12-month observation period among Medicare fee-for-service long-stay residents (in a NH >=90 days) who are >=65 years old and who have NEITHER advanced dementia NOR advanced congestive heart failure/chronic obstructive lung disease
Time Frame: 12-month observation period
Measure: Mean (Standard Deviation); unit: person-years
Arm/Group | ACP Video Program | Usual ACP Procedures
Number analyzed (Participants) | 5766 | 11782
person-years | 1.65 (3.9) | 1.68 (4.8)

3. Secondary Outcome: Hospital Transfer Rate Among Short-stay Residents With Advanced Illness
Description: Number of hospital transfers (number of transfers/person-days alive) over a 100-day observation period among Medicare fee-for-service short-stay residents (in a NH <90 days) who are >=65 years old and who have EITHER advanced dementia OR advanced congestive heart failure/chronic obstructive lung disease
Time Frame: 100-day observation period
Measure: Mean (Standard Deviation); unit: person-years
Arm/Group | ACP Video Program | Usual ACP Procedures
Number analyzed (Participants) | 2538 | 5290
person-years | 6.9 (17.8) | 6.8 (16.8)

4. Secondary Outcome: Hospital Transfer Rate Among Short-stay Residents Without Advanced Illness
Description: Number of hospital transfers (number of transfers/person-days alive) over a 100-day observation period among Medicare fee-for-service short-stay residents (in a NH <90 days) who are >=65 years old and who have NEITHER advanced dementia NOR advanced congestive heart failure/chronic obstructive lung disease
Time Frame: 100-day observation period
Measure: Mean (Standard Deviation); unit: person-years
Arm/Group | ACP Video Program | Usual ACP Procedures
Number analyzed (Participants) | 23304 | 50195
person-years | 4.5 (10.3) | 4.4 (10.4)

5. Secondary Outcome: Proportion of Target Cohort With Last Observed Advance Directive Status
Description: Proportion of long-stay residents (in a NH >=90 days) who are >=65 years old and who have EITHER advanced dementia OR advanced congestive heart failure/chronic obstructive lung disease whose last observed advance directive status during their 12-month observation period was: Full Code, Do Not Resuscitate (NOT Do Not Hospitalize), or Do Not Hospitalize. A resident whose last observed status was both Do Not Resuscitate and Do Not Hospitalize is categorized as Do Not Hospitalize only. Analyses will be limited to Genesis HealthCare facilities in which >75% of residents have any advance directive because the remaining Genesis HealthCare and PruittHealth facilities do not have reliable sources for these data.
Time Frame: 12-month observation period
Measure: Count of Participants; unit: Participants
Arm/Group | Advance Care Planning (ACP) Video Program | Usual Advance Care Planning (ACP) Procedures
Number analyzed (Participants) | 1970 | 2880
Participants
  Full Code | 295 | 570
  Do Not Resuscitate | 1288 | 2010
  Do Not Hospitalize | 387 | 300

6. Secondary Outcome: Proportion of Long-stay Residents Without Advanced Illness With Last Observed Advance Directive Status
Description: Proportion of long-stay residents (in a NH >=90 days) who are >=65 years old and who do have NEITHER advanced dementia NOR advanced congestive heart failure/chronic obstructive lung disease whose last observed advance directive status during their 12-month observation period was: Full Code, Do Not Resuscitate (NOT Do Not Hospitalize), or Do Not Hospitalize. A resident whose last observed status was both Do Not Resuscitate and Do Not Hospitalize is categorized as Do Not Hospitalize only. Analyses will be limited to Genesis HealthCare facilities in which >75% of residents have any advance directive because the remaining Genesis HealthCare and PruittHealth facilities do not have reliable sources for these data.
Time Frame: 12-month observation period
Measure: Count of Participants; unit: Participants
Arm/Group | Advance Care Planning (ACP) Video Program | Usual Advance Care Planning (ACP) Procedures
Number analyzed (Participants) | 3233 | 5659
Participants
  Full Code | 1150 | 2210
  Do Not Resuscitate | 1714 | 3018
  Do Not Hospitalize | 369 | 431

7. Secondary Outcome: Proportion of Short-stay Residents With Advanced Illness With Last Observed Advance Directive Status
Description: Proportion of short-stay residents (in a NH <90 days) who are >=65 years old and who have EITHER advanced dementia OR advanced congestive heart failure/chronic obstructive lung disease whose last observed advance directive status during their 100-day observation period was: Full Code, Do Not Resuscitate (NOT Do Not Hospitalize), or Do Not Hospitalize. A resident whose last observed status was both Do Not Resuscitate and Do Not Hospitalize is categorized as Do Not Hospitalize only. Analyses will be limited to Genesis HealthCare facilities in which >75% of residents have any advance directive because the remaining Genesis HealthCare and PruittHealth facilities do not have reliable sources for these data.
Time Frame: 100-day observation period
Measure: Count of Participants; unit: Participants
Arm/Group | Advance Care Planning (ACP) Video Program | Usual Advance Care Planning (ACP) Procedures
Number analyzed (Participants) | 1166 | 1701
Participants
  Full Code | 482 | 761
  Do Not Resuscitate | 581 | 858
  Do Not Hospitalize | 103 | 82

8. Secondary Outcome: Proportion of Short-stay Residents Without Advanced Illness With Last Observed Advance Directive Status
Description: Proportion of short-stay residents (in a NH <90 days) who are >=65 years old and who have NEITHER advanced dementia NOR advanced congestive heart failure/chronic obstructive lung disease whose last observed advance directive status during their 100-day observation period was: Full Code, Do Not Resuscitate (NOT Do Not Hospitalize), or Do Not Hospitalize. A resident whose last observed status was both Do Not Resuscitate and Do Not Hospitalize is categorized as Do Not Hospitalize only. Analyses will be limited to Genesis HealthCare facilities in which >75% of residents have any advance directive because the remaining Genesis HealthCare and PruittHealth facilities do not have reliable sources for these data.
Time Frame: 100-day observation period
Measure: Count of Participants; unit: Participants
Arm/Group | Advance Care Planning (ACP) Video Program | Usual Advance Care Planning (ACP) Procedures
Number analyzed (Participants) | 13292 | 19784
Participants
  Full Code | 8289 | 12899
  Do Not Resuscitate | 4541 | 6392
  Do Not Hospitalize | 462 | 493

9. Secondary Outcome: Proportion of Target Cohort Receiving Any Burdensome Treatment
Description: Proportion of long-stay residents (in a NH >=90 days) who are >=65 years old and who have EITHER advanced dementia OR advanced congestive heart failure/chronic obstructive lung disease who receive any burdensome treatment (new feeding tube insertions, parenteral therapy, intubation, ICU care) during a 12-month observation period
Time Frame: 12-month observation period
Measure: Count of Participants; unit: Participants
Arm/Group | ACP Video Program | Usual ACP Procedures
Number analyzed (Participants) | 4171 | 8308
Participants | 453 | 971

10. Secondary Outcome: Proportion of Long-stay Residents Without Advanced Illness Receiving Any Burdensome Treatment
Description: Proportion of long-stay residents (in a NH >=90 days) who are >=65 years old and who have NEITHER advanced dementia NOR advanced congestive heart failure/chronic obstructive lung disease who receive any burdensome treatment (new feeding tube insertions, parenteral therapy, intubation, ICU care) during a 12-month observation period
Time Frame: 12-month observation period
Measure: Count of Participants; unit: Participants
Arm/Group | ACP Video Program | Usual ACP Procedures
Number analyzed (Participants) | 5766 | 11782
Participants | 465 | 1028

11. Secondary Outcome: Proportion of Short-stay Residents With Advanced Illness Receiving Any Burdensome Treatment
Description: Proportion of short-stay residents (in a NH <90 days) who are >=65 years old and who have EITHER advanced dementia OR advanced congestive heart failure/chronic obstructive lung disease who receive any burdensome treatment (new feeding tube insertions, parenteral therapy, intubation, ICU care) during a 100-day observation period among
Time Frame: 100-day observation period
Measure: Count of Participants; unit: Participants
Arm/Group | ACP Video Program | Usual ACP Procedures
Number analyzed (Participants) | 2538 | 5290
Participants | 294 | 621

12. Secondary Outcome: Proportion of Short-stay Residents Without Advanced Illness Receiving Any Burdensome Treatment
Description: Proportion of short-stay residents (in a NH <90 days) who are >=65 years old and who have NEITHER advanced dementia NOR advanced congestive heart failure/chronic obstructive lung disease who receive any burdensome treatment (new feeding tube insertions, parenteral therapy, intubation, ICU care) during a 100-day observation period
Time Frame: 100-day observation period
Measure: Count of Participants; unit: Participants
Arm/Group | ACP Video Program | Usual ACP Procedures
Number analyzed (Participants) | 23304 | 50195
Participants | 1726 | 3405

13. Secondary Outcome: Proportion of Target Cohort With Any Hospice Enrollment
Description: Proportion of long-stay residents (in a NH >=90 days) who are >=65 years old and who have EITHER advanced dementia OR advanced congestive heart failure/chronic obstructive lung disease with any hospice enrollment during a 12-month observation period
Time Frame: 12-month observation period
Measure: Count of Participants; unit: Participants
Arm/Group | ACP Video Program | Usual ACP Procedures
Number analyzed (Participants) | 4171 | 8308
Participants | 904 | 1878

14. Secondary Outcome: Proportion of Long-stay Residents Without Advanced Illness With Any Hospice Enrollment
Description: Proportion of long-stay residents (in a NH >=90 days) who are >=65 years old and who have NEITHER advanced dementia NOR advanced congestive heart failure/chronic obstructive lung disease with any hospice enrollment during a 12-month observation period
Time Frame: 12-month observation period
Measure: Count of Participants; unit: Participants
Arm/Group | ACP Video Program | Usual ACP Procedures
Number analyzed (Participants) | 5766 | 11782
Participants | 373 | 832

15. Secondary Outcome: Proportion of Short-stay Residents With Advanced Illness With Any Hospice Enrollment
Description: Proportion of short-stay residents (in a NH <90 days) who are >=65 years old and who have EITHER advanced dementia OR advanced congestive heart failure/chronic obstructive lung disease with any hospice enrollment during a 100-day observation period
Time Frame: 100-day observation period
Measure: Count of Participants; unit: Participants
Arm/Group | ACP Video Program | Usual ACP Procedures
Number analyzed (Participants) | 2538 | 5290
Participants | 588 | 1220

16. Secondary Outcome: Proportion of Short-stay Residents Without Advanced Illness With Any Hospice Enrollment
Description: Proportion of short-stay residents (in a NH <90 days) who are >=65 years old and who have NEITHER advanced dementia NOR advanced congestive heart failure/chronic obstructive lung disease with any hospice enrollment during a 100-day observation period
Time Frame: 100-day observation period
Measure: Count of Participants; unit: Participants
Arm/Group | ACP Video Program | Usual ACP Procedures
Number analyzed (Participants) | 23304 | 50195
Participants | 2273 | 4875

17. Secondary Outcome: Proportion of Target Cohort That Has Medicare ACP Billing Codes
Description: Proportion of long-stay residents (in a NH >=90 days) who are >=65 years old and who have EITHER advanced dementia OR advanced congestive heart failure/chronic obstructive lung disease who have any Medicare ACP billing code during their 12-month observation period
Time Frame: 12-month observation period
Measure: Count of Participants; unit: Participants
Arm/Group | ACP Video Program | Usual ACP Procedures
Number analyzed (Participants) | 4171 | 8308
Participants | 356 | 685

18. Secondary Outcome: Proportion of Long-stay Residents Without Advanced Illness That Has Medicare ACP Billing Codes
Description: Proportion of long-stay residents (in a NH >=90 days) who are >=65 years old and who have NEITHER advanced dementia NOR advanced congestive heart failure/chronic obstructive lung disease who have any Medicare ACP billing code during their 12-month observation period
Time Frame: 12-month observation period
Measure: Count of Participants; unit: Participants
Arm/Group | ACP Video Program | Usual ACP Procedures
Number analyzed (Participants) | 5766 | 11782
Participants | 571 | 1157

19. Secondary Outcome: Proportion of Short-stay Residents With Advanced Illness That Has Medicare ACP Billing Codes
Description: Proportion of short-stay residents (in a NH <90 days) who are >=65 years old and who have EITHER advanced dementia OR advanced congestive heart failure/chronic obstructive lung disease who have any Medicare ACP billing code during their 100-day observation period
Time Frame: 100-day observation period
Measure: Count of Participants; unit: Participants
Arm/Group | ACP Video Program | Usual ACP Procedures
Number analyzed (Participants) | 2538 | 5290
Participants | 224 | 479

20. Secondary Outcome: Proportion of Short-stay Residents Without Advanced Illness That Has Medicare ACP Billing Codes
Description: Proportion of short-stay residents (in a NH <90 days) who are >=65 years old and who have NEITHER advanced dementia NOR advanced congestive heart failure/chronic obstructive lung disease who have any Medicare ACP billing code during their 100-day observation period
Time Frame: 100-day observation period
Measure: Count of Participants; unit: Participants
Arm/Group | ACP Video Program | Usual ACP Procedures
Number analyzed (Participants) | 23304 | 50195
Participants | 1669 | 4068

ADVERSE EVENTS:
Time Frame: 12 months
Description: We had three mechanisms to capture potential serious adverse events: (1) 'Serious Negative Reaction' Form and protocol to be initiated by nursing home staff within 4 hours of an observed event; (2) Entry of observed event details by nursing home staff in a Video Status Report User-Defined Assessment (VSR UDA) embedded in the electronic medical record system; and (3) Qualitative interviews conducted by research staff with nursing home staff that included questions about observed events.
Arm/Group | ACP Video Program | Usual ACP Procedures
All-Cause Mortality (participants affected / at risk) | 8403/33035 | 17251/70013
Serious Adverse Events (participants affected / at risk) | 0/33035 | 0/70013
Other Adverse Events (participants affected / at risk) | 0/33035 | 0/70013

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-17): https://cdn.clinicaltrials.gov/large-docs/88/NCT02612688/Prot_SAP_000.pdf